Official title of the study :Efficacy of Oral Bovine Lactoferrin on Prevention of Neonatal Sepsis, Necrotizing Enterocolitis and its effect on CBC in Preterm infants. (stastical analysis)

Date of document 1 June 2019

#### **Results**

The results of the the current study are presented in the following tables and figures:-



NEC = necrotizing enterocolitis, BPD= bronchopulmonary dysplasia RDS = respiratory distress syndrome

Figure (7): Consort flow chart of studied preterm neonates

Table (13): Demographic data of placebo group and once daily lactoferrin supplemented group:-

| Personal ( | Personal data | | cebo<br>oup<br>100) | da<br>gre | nce<br>nily<br>oup<br>100) | Test<br>valu<br>e | P. value |
|---|---|---|---|---|---|---|---|
| | | No<br>· | % | No . | % | | |
| | Nearterm (34-<br>36) | 35 | 35.<br>0 | 35 | 35.<br>0 | | |
| GA preterm (in weeks) | Moderate (32-33) | 40 | 40.<br>0 | 40 | 40.<br>0 | 0.225 | 0.614 |
| weeks) | Severe (28-31) | 22 | 22.<br>0 | 22 | 22.<br>0 | | |
| | Extreme (<28) | 3 | 3.0 | 3 | 3.0 | | |
| GA (weeks) | Mean±SD | 30.47±2. | | | 6±2.<br>7 | 1.42 | 0.156 |
| | Range | 26 - 36 | | 26 - 36 | | | |
| Sex | Male | 64 | 64.<br>0 | 53 | 53.<br>0 | 2.06 | 0.151 |
| | Female | 36 | 36.<br>0 | 47 | 47.<br>0 | 0 | 0.131 |
| | First | 15 | 15.<br>0 | 20 | 20.<br>0 | | 0.258 |
| Order of birth | Second | 20 | 20.<br>0 | 22 | 22.<br>0 | 4.03 | |
| Order of birth | Third | 31 | 31.<br>0 | 19 | 19.<br>0 | 2 | 0.238 |
| | >third | 34 | 34.<br>0 | 39 | 39.<br>0 | | |
| | Single | 72 | 72.<br>0 | 61 | 61.<br>0 | 2.24 | |
| Single/Multiple birth | Twins | 28 | 28.<br>0 | 39 | 39.<br>0 | 4 | 0.105 |
| | Triple | 0 | 0.0 | 0 | 0.0 | | |
| Mode of delivery | NVD | 65 | 65.<br>0 | 54 | 54.<br>0 | 2.07 | 0.150 |
| Mode of delivery | CS | 35 35. 46 46. | | 46.<br>0 | 5 | 0.130 | |
| Apgar 1 minute | Median(IQR) | 8(7 | 7-9) | 8(7 | 7-9) | 6.39<br>4 | 0.371 |

| Apgar 5 minute | Median(IQR) | 9(9-10) | 9(9-10) | 0.95<br>9 | 0.690 |
|----------------|-------------|---------|---------|-----------|-------|
|----------------|-------------|---------|---------|-----------|-------|

As regards demographic data, there were no significant statistical difference between placebo and oral lactoferrin groups.

Table (14): Comparison between placebo group and once daily lactoferrin supplemented group regarding maternal and obstetric data:

| Maternal history | | | Placebo<br>(n=100) | | Lactoferri<br>n (n=100) | | P.<br>value |
|---|---|---|---|---|---|---|---|
| | | | % | No. | % | | |
| Maternal Age (years) | Mean±S<br>D | 28.65 | 28.65±6.52 | | 8±6.67 | 1.64 | 0.102 |
| | Range | 19 - 47 | | 19 - 45 | | | |
| Maternal DM | Positive | 8 | 8.0 | 12 | 12.0 | 0.50 | 0.050 |
| Maternal DM | Negative | 92 | 92.0 | 88 | 88.0 | 0 | 0.030 |
| Maternal HTN | Positive | 11 | 11.0 | 14 | 14.0 | 0.18 | 0.669 |
| Maternal H I N | Negative | 89 | 89.0 | 86 | 86.0 | 3 | 0.009 |
| Anti partum | Positive | 3 | 3.0 | 14 | 14.0 | 6.42 | 0.011 |
| Hemorrhage | Negative | 97 | 97.0 | 86 | 86.0 | 9 | * |

Independent samples T Test and Chi-square test

This table shows that there is significant statistical higher incidence of anti-partum hemorrhage among placebo group than in oral lactoferrin supplemented group.

<sup>\*</sup> Statistically significant difference (p<0.05)

<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

<sup>\*</sup> Statistically significant difference (p<0.05)

<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

Table (15):- Comparison between placebo group and once daily lactoferrin supplemented group as regarding anthropometric measures and vital data upon admission:

| | Examination on admission | | Placebo<br>group<br>(n=100) | | e daily<br>oup<br>(100) | Test<br>valu | P.<br>value |
|---|---|---|---|---|---|---|---|
| dumiss | 51011 | No | % | No. | % | е | varac |
| Birth weight | 5th - 95<br>th | 90 | 90.0 | 88 | 88.0 | 0.82 | 0.662 |
| (on centile) | <5th | 5 | 5.0 | 8 | 8.0 | 6 | 0.662 |
| | >95th | 5 | 5.0 | 4 | 4.0 | | |
| Birth weight (kilogram) | Mean±S<br>D | 1.55±0.55 | | 1.45±0.45 | | 1.062 | 0.29 |
| Length at | 5th - 95<br>th | 87 | 87.0 | 90 | 90.0 | 0.47 | 0.69 |
| birth (on | <5th | 7 | 7.0 | 5 | 5.0 | 5 | |
| centile) | >95th | 6 | 6.0 | 5 | 5.0 | | |
| Length at birth | Mean±S<br>D | 42. | 20±3.<br>6 | 40.1 | 1±3.7 | 2.94 | 0. 64 |
| (Centimeter) | Range | 36 | 5 - 48 | 36 | - 48 | 0 | |
| Head | 5th - 95<br>th | 98 | 98.0 | 98 | 98.0 | 0.22 | 0.614 |
| circumferanc | <5th | 2 | 2.0 | 2 | 2.0 | 5 | 0.614 |
| e (on centile) | >95th | 0 | 0.0 | 0 | 0.0 | | |
| Head | Mean±S | 30. | 40±1. | 30.5 | 0±1.8 | 1.28 | 0.202 |

| circumferanc | D | 75 | 5 | | |
|---|---|---|---|---|---|
| e<br>(Centimeter) | Range | 26 - 34 | 26 - 34 | 1 | |
| Tomoroturo | Mean±S<br>D | 36.30±0.<br>30 | 36.40±0.4<br>0 | 0.28 | 0.773 |
| Temperature | Range | 36.8 -<br>37.2 | 36.8 - 37.1 | 9 | 0.775 |
| Heart rate | Mean±S<br>D | 120.8±14<br>.2 | 118.6±16.<br>68 | 1.31 | 0.189 |
| | Range | 80 - 146 | 86 - 154 | 0 | |
| Respiratory | Mean±S<br>D | 48.3±10.<br>80 | 46.5±10.4 | 0.48 | 0.628 |
| rate | Range | 36 - 62 | 34 - 64 | 5 | |
| Systolic blood | Mean±S<br>D | 62.2±6.2 | 62.6±7.8 | 0.52 | 0.601 |
| pressure | Range | 48 - 78 | 46 - 78 | 4 | |
| Diastolic<br>blood | Mean±S<br>D | 38.4±8.6 | 36.6±7.6 | 0.60 | 0.546 |
| pressure | Range | 26 - 50 | 26 - 52 | 4 | |

The table shows that there was non significant statistical difference between placebo group and once daily lactoferrin supplemented group as regarding anthropometric measures and vital signs.

<sup>\*</sup> Statistically significant difference (p<0.05)

<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

Table (16): Comparison between placebo group and once daily lactoferrin supplemented group regarding development of clinical signs of sepsis according to Tollner score:

| | | gr | cebo<br>oup<br>:100) | da<br>gr | nce<br>aily<br>oup<br>100) | Test<br>valu<br>e | P. value |
|---|---|---|---|---|---|---|---|
| | | No | % | No | % | | |
| | Normal | 84 | 84.<br>0 | 92 | 92.<br>0 | | |
| Skin color | Moderate change | 7 | 7.0 | 8 | 8.0 | 9.43<br>0 | 0.009** |
| | Sever<br>change | 9 | 9.0 | 0 | 0.0 | | |
| Temp | Positive | 13 | 13.<br>0 | 6 | 6.0 | 2.09 | 0.148 |
| instability | Negative | 87 | 87.<br>0 | 94 | 94.<br>0 | 4 | 0.140 |
| Respiratory<br>signs O2<br>requirement | Normal | 59 | 59.<br>0 | 54 | 54.<br>0 | | |
| | 02 | 18 | 18.<br>0 | 26 | 26.<br>0 | 8.58 | 0.035 |
| | СРАР | 10 | 10.<br>0 | 8 | 8.0 | 3 | 0.033 |
| | IMV | 13 | 13.<br>0 | 12 | 12.<br>0 | | |
| Apnea | Positive | 18 | 18.<br>0 | 10 | 10.<br>0 | 2.03 | 0.154 |
| Арпса | Negative | 82 | 82.<br>0 | 90 | 90.<br>0 | 5 | 0.154 |
| Inter and subcostal | Positive | 36 | 36.<br>0 | 30 | 30.<br>0 | 0.56 | 0.452 |
| retraction | Negative | 64 | 64.<br>0 | 70 | 70.<br>0 | 5 | 0.432 |
| Teachypnea | Positive | 34 | 34.<br>0 | 30 | 30.<br>0 | 0.20 | 0.650 |
| icacitypilea | Negative | 66 | 66.<br>0 | 70 | 70.<br>0 | 7 | 0.030 |
| Cyanosis | Positive | 13 | 13.<br>0 | 10 | 10.<br>0 | 0.19 | 0.658 |
| Cyanosis | Negative | 87 | 87.<br>0 | 90 | 90.<br>0 | 7 | 0.038 |
| Grunting | Positive | 18 | 18.<br>0 | 11 | 11.<br>0 | 1.45<br>2 | 0.228 |

| | | gr | cebo<br>oup<br>:100) | da<br>gr | nce<br>aily<br>oup<br>:100) | Test<br>valu<br>e | P. value |
|---|---|---|---|---|---|---|---|
| | | No | % | No | % | | |
| | Negative | 82 | 82.<br>0 | 89 | 89.<br>0 | | |
| Circulatory signs | Positive | 12 | 12.<br>0 | 10 | 10.<br>0 | 0.05 | 0.820 |
| Bradycardia | Negative | 88 | 88.<br>0 | 90 | 90.<br>0 | 1 | |
| Weak pulse | Positive | 14 | 14.<br>0 | 9 | 9.0 | 33.7 | <0.001* |
| weak puise | Negative | 86 | 86.<br>0 | 91 | 91.<br>0 | 45 | * |
| | Positive | 6 | 6.0 | 2 | 2.0 | 0.20 | |
| Shock | Negative | 94 | 94.<br>0 | 98 | 98.<br>0 | 7 | 0.650 |
| | Normal | 80 | 80.<br>0 | 92 | 92.<br>0 | | |
| CFT | Impaired | 11 | 11.<br>0 | 2 | 2.0 | 7.67<br>0 | 0.022* |
| | Considerab<br>ly impaired | 9 | 9.0 | 6 | 6.0 | | |
| Hypotension | Positive | 11 | 11.<br>0 | 7 | 7.0 | 0.54 | 0.459 |
| Пуросензіон | Negative | 89 | 89.<br>0 | 93 | 93.<br>0 | 9 | 0.439 |
| GIT signs<br>Abdominal | Positive | 16 | 16.<br>0 | 7 | 7.0 | 3.14 | 0.076 |
| distension | Negative | 84 | 84.<br>0 | 93 | 93.<br>0 | 4 | 0.076 |
| Feeding | Positive | 31 | 31.<br>0 | 12 | 12.<br>0 | 9.60 | 0.002** |
| intolerance | Negative | 69 | 69.<br>0 | 88 | 88.<br>0 | 0 | 0.002 |
| Diarrhea | Positive | 22 | 22.<br>0 | 8 | 8.0 | 6.62 | 0.010* |
| Diaiiilea | Negative | 78 | 78.<br>0 | 92 | 92.<br>0 | 7 | 0.010. |
| Henatomogaly | 0 - 2 cm | 83 | 83.<br>0 | 94 | 94.<br>0 | 9.96 | 0.007** |
| Hepatomegaly | 2 - 4 cm | 8 | 8.0 | 6 | 6.0 | 9 | 0.007 |
| | >4 cm | 9 | 9.0 | 0 | 0.0 | | |
| <b>D</b> | Positive | 3 | 3.0 | 0 | 0.0 | 1.48 | 0.000 |
| Bloody stool | Negative | 97 | 97.<br>0 | 10<br>0 | 100<br>.0 | 4 | 0.223 |

| | | gr | cebo<br>oup<br>:100) | di<br>gr | nce<br>aily<br>oup<br>:100) | Test<br>valu<br>e | P. value |
|---|---|---|---|---|---|---|---|
| | | No | % | No | % | | |
| Jaundice | Positive | 23 | 23.<br>0 | 8 | 8.0 | 7.48 | .006** |
| Jadridice | Negative | 77 | 77.<br>0 | 92 | 92.<br>0 | 2 | .000 |
| Neurological | Positive | 8 | 8.0 | 4 | 4.0 | 0.79 | |
| signs Irritbility | Negative | 92 | 92.<br>0 | 96 | 96.<br>0 | 8 | 0.372 |
| | Normal | 74 | 74.<br>0 | 98 | 98.<br>0 | | |
| Hypotonia | Hypotonia | 13 | 13.<br>0 | 2 | 2.0 | 24.4<br>16 | <0.001* |
| | Floppy | 13 | 13.<br>0 | 0 | 0.0 | | |
| W.B.C count | Normal<br>Leucocytos<br>is<br>Leucopenia | 82<br>18<br>0 | 82.<br>0<br>18.<br>0<br>0.0 | 95<br>5<br>0 | 95.<br>0<br>5.0<br>0.0 | 8.97<br>1 | 0.012* |
| Shift to left | No<br>Moderate<br>severe | 82<br>10<br>8 | 82.<br>0<br>10.<br>0<br>8.0 | 95<br>4<br>1 | 95.<br>0<br>4.0<br>1.0 | 8.97<br>1 | 0.012* |
| | Normal | 90 | 90.<br>0 | 94 | 94.<br>0 | | |
| Others blood glucose level | Hypoglyce<br>mia | 3 | 3.0 | 2 | 2.0 | 1.10<br>5 | 0.576 |
| | Hyperglyce<br>mia | 7 | 7.0 | 4 | 4.0 | | |
| D | Positive | 6 | 6.0 | 2 | 2.0 | 1.17 | 0.270 |
| Petechiae | Negative | 94 | 94. | 98 | 98. | 2 | 0.279 |
| Thrombocytop<br>enia | Positive<br>Negative | 96 | 96.<br>0 | 99 | 99.<br>0 | 0.00 | 0.959 |
| | Positive | 0 | 0.0 | 0 | 0.0 | 0.00 | |
| DIC | Negative | 10<br>0 | 100 | 10<br>0 | 100.<br>0 | 0.00 | 0.000 |
| Oral fungal | Positive | 16 | 16.<br>0 | 3 | 3.0 | 7.97 | 005** |
| infection | Negative | 84 | 84.<br>0 | 97 | 97.<br>0 | 7 | .005** |

| | | gr | cebo<br>oup<br>:100) | Once<br>daily<br>group<br>(n=100) | | Test<br>valu<br>e | P. value |
|---|---|---|---|---|---|---|---|
| | | No | % | No | % | | |
| | No sepsis | 82 | 82.<br>0 | 95 | 95.<br>0 | | 0.012* |
| Tollner score | Observatio<br>n range | 10 | 10.<br>0 | 4 | 4.0 | 8.97<br>1 | |
| | Suspicison of sepsis | 8 | 8.0 | 1 | 1.0 | | |

The table shows that oral lactoferrin supplemented group had significant lower Tollner score (signs of sepsis) compared with placebo group.

Figure (8): Tollner score among the two groups



Showing that there is significant lower incidence of sepsis in lactoferrin supplemented group in comparison with placebo group.

<sup>\*</sup> Statistically significant difference (p<0.05)

<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

| Other investigations | | Placebo group (n=100) | | Once d<br>(n=100 | laily group | Test<br>value | P. valu |
|---|---|---|---|---|---|---|---|
| | | No. | % | No. | % | | |
| Hb on admission (g/dl) | Mean±S<br>D | 14.56±4.52 | | 14.44± | 14.44±3.41 | | 0.321 |
| | Range | 10.40 - 19.5 | | 10.4 - | 10.4 - 19.8 | | |
| CRP on admission | Negative | 100 | 100.0 | 100 | 100 | 58.851 | 1.00 |
| CKF on admission | Positive | 0 | 0.0 | 0 | 0.0 | 30.031 | |
| CRP in follow up (who | Negative | 82 | 82.0 | 95 | 95.0 | 17.960 | 0.008* |
| develop sepsis) | Positive | 18 | 18.0 | 5 | 5 | 17.869 | |

# Table (17): Comparison between placebo group and once daily lactoferrin supplemented group regarding hemoglobin and CRP.

HB = hemoglobin, CRP = c-reactive protein

Independent samples T Test and Chi-square test

\* Statistically significant difference (p<0.05)

\*\*Highly statistically significant difference (p<0.01)

This table shows that there was a significantly lower incidence of positive CRP in oral lactoferrin supplemented group than in placebo one (during follow up)

Figure (9) Comparison between placebo group and once daily lactoferrin supplemented group regarding CRP



This figure shows that positive CRP is significant statistically higher in placebo group than in lactoferrin supplemented one during follow up.

Table (18) comparison between placebo and oral supplemented groups regarding ALT,AST and billirubin.

| | Placebo | Lactoferrin | Test | Р |
|------------|--------------|--------------|-------|------|
| | group | | value | valu |
| | | | | e |
| ALT (U\L) | 28.77±6.30 | 28.14±5.26 | 0.272 | 0.87 |
| at one | | | | 6 |
| month | | | | |
| AST (U\L) | 37.55±5.31 | 38.22±4.23 | 2.876 | 0.06 |
| at one | | | | 7 |
| month | | | | |
| Billirubin | 3.4(2.2-5.3) | 3.5(2.6-5.2) | 3.367 | 0.09 |
| (mg\dl) at | | | | 2 |
| one month | | | | |

ALT= alanine transaminase , AST= aspartate aminotransferase

Independent samples T Test and Chi-square test

This table shows no signifificant statistical difference between ALT , AST and billirubin in the two studied groups.

Table(19): Comparison between placebo group and once daily lactoferrin supplemented group as regard arterial blood gases on admission and during sepsis:

| ABG on admission | | Placebo group<br>(n=100) | lactoferrin group<br>(n=100) | Test<br>value | P. value |
|---|---|---|---|---|---|
| PH | Mean±SD | 7.36±0.0812 | 7.37±0.0735 | 0.246 | 0.624 |
| rn | Range | 7.28 - 7.44 | 7.27 - 7.46 | 0.246 | 0.024 |

<sup>\*</sup> Statistically significant difference (p<0.05)

<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

#### Results

| Pco2 | Mean±SD | 37.22±9.99 | 37.24±10.44 | 0.242 | 0.816 |
|---|---|---|---|---|---|
| PC02 | Range | 17 - 68.5 | 19 - 60.2 | 0.242 | 0.810 |
| BD | Mean±SD | -4.12±6.88 | -4.81±6.98 | 0.237 | 0.457 |
| Dυ | Range | -9 - 3.1 | -8.8 - 3.6 | 0.237 | 0.437 |
| Hco3 | Mean±SD | 18.46±5.9 | 18.88±5.4 | 0.345 | 0.534 |
| псоз | Range | 13.5 - 25.4 | 13.2 - 25.3 | 0.343 | 0.554 |
| ADC 1 | | Placebo group | Lactoferrin group | Test | D volvo |
| ABG during se | DSIS | (n=100) | (n=100) | value | P. value |
| PH | Mean±SD | 7.30±0.26 | 7.36±0.07 | 3.748 | <0.001** |
| rn | Range | 7.14 - 7.42 | 7.33 - 7.37 | 3.748 | <0.001 |
| Pco2 | Mean±SD | 34.43±8.32 | 30.3±8.1 | 7.030 | <0.001** |
| PC02 | Range | 24 - 52 | 20.1 - 38.7 | 7.030 | <0.001 |
| BD | Mean±SD | -6.98±5.66 | -6.41±4.3 | 3.094 | .002** |
| DD | Danas | -13.1 - 6.7 | -8.12.6 | 3.094 | .002 |
| | Range | -13.1 - 0.7 | -0.12.0 | | |
| Hco3 | Mean±SD | 17.54±3.82 | 18.15±3.62 | 0.589 | 0.557 |

BD=base deficit

Independent samples T Test

This table shows that upon development of sepsis lactoferrin supplemented group has a higher PH and lower BD compared with oral placebo group.

Table (20): Lab analysis on day7

| Variable | Lactoferrin<br>(n=100) | Placeho (n=100) | | P.<br>value |
|---|---|---|---|---|
| | Mean±SD | Mean±SD | value | value |
| Serum ferritin (ng/ml) | 332.4±43.2 | 338.7±55.2 | 1.855 | 0.065 |
| Hemoglobin (g/dl) | 15.8±2.9 | 15.3±2.4 | 4.359 | 0.078 |
| Hematocrit (%) | 45.1±6.6 | 42.2±6.3 | 4.659 | 0.064 |
| MCV (fl) | 100.1±4.4 | 97.3±8.2 | 3.200 | 0.063 |

<sup>\*</sup> Statistically significant difference (p<0.05)

<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

| RDW (%) | 17.2±2.3 | 17.1±3.2 | 0.966 | 0.335 |
|---|---|---|---|---|
| Platelets (x1, 000/mm <sup>3</sup> ) | 175.4±73.2 | 178.3±100.3 | 0.890 | 0.374 |
| TLC (x1, 000/mm <sup>3</sup> ) | 13.4±5.2 | 12.8±5.4 | 1.106 | 0.270 |

Data are mean  $\pm$  SD or number (%)

Independent samples T Testand Chi-square test

MCV = mean corpuscular volume ,RDW= red cell distribution widths , PLT=platelets , TLC = total leucocytic count.

There was no stastically significant difference between the 2 groups as regards S.ferritin, hemoglobin, hematocrit, MCV, RDW, platelets and TLC on day 7.

Table (21): Lab analysis on day30

| Variable | Lactoferrin<br>(n=100) | Placebo<br>(n=100) | Test<br>value | P. value |
|---|---|---|---|---|
| | Mean±SD | Mean±SD | | |
| Serum ferritin (ng/ml) | 377.9±68.6 | 290.7±70.9 | 11.61 | <0.001** |
| Hemoglobin (g/dl) | 15.1±1.9 | 11.3±2.2 | 5.243 | <0.001** |
| Hematocrit (%) | 47.4±3.5 | 38.1±6.9 | 11.64 | <0.001** |

<sup>\*</sup> Statistically significant difference (p<0.05).

<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

| | | | 7 | |
|---|---|---|---|---|
| MCV (fl) | 99.9±4.8 | 90.3±8.5 | 7.417 | <0.001** |
| RDW (%) | 15.9±1.6 | 17.8±2.9 | 4.226 | <0.001** |
| Platelets (x1, 000/mm <sup>3</sup> ) | 248.3±64.4 | 252.1±140.2 | 0.461 | 0.645 |
| TLC (x1, 000/mm <sup>3</sup> ) | 13.1±3.1 | $17.4 \pm 8.1$ | 6.145 | <0.001* |

MCV = mean corpuscular volume , RDW = red cell distribution widths PLT=platelets , TLC = total leucocytic count .

The lactoferrin group showed statistically significant higher S.ferritin level ,HB ,HCT,MCV than placebo supplemented group

But lactoferrin group showed significant statistical lower RDW, and TLC .

NO statistical difference for PLT count.

Table (22):Comparison between day 7 and 30 in each group as regards S.ferritin ,Hb, HCT, MCV,RDW, PLT and TLC.

| Grou | Variable | Time | Mean | SD | P. value |
|------|----------|------|------|----|----------|
| p | | | | | |

<sup>\*</sup> Statistically significant difference (p<0.05)

<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

| | G C '4' ( / D) | Day 7 | 332.4 | 43.2 | <0.001* |
|---|---|---|---|---|---|
| | Serum ferritin (ng/ml) | Day 30 | 377.9 | 68.6 | * |
| | Hamadakir (a/dl) | Day 7 | 15.8 | 2.9 | 0.0694 |
| Lactoferrin (n=100) | Hemoglobin (g/dl) | Day 30 | 15.1 | 1.9 | 0.0684 |
| | Homotoppit (9/) | Day 7 | 45.1 | 6.6 | 0.375 |
| <b> </b> | Hematocrit (%) | Day 30 | 47.4 | 3.5 | 0.373 |
| <u> </u> | MCV (4) | Day 7 | 100.1 | 4.4 | 0.682 |
| | MCV (fl) | Day 30 | 99.9 | 4.8 | 0.082 |
| ofe | RDW (%) | Day 7 | 17.2 | 2.3 | 0.001** |
| | KD W (78) | Day 30 | 15.9 | 1.6 | 0.001 |
| | Platelets (x1, 000/mm <sup>3</sup> ) | Day 7 | 175.4 | 73.2 | <0.001* |
| | | Day 30 | 248.3 | 64.4 | * |
| | TLC (x1, 000/mm <sup>3</sup> ) | Day 7 | 13.4 | 5.2 | 0.191 |
| | | Day 30 | 13.1 | 3.1 | 0.191 |
| | Serum ferritin (ng/ml) | Day 7 | 338.7 | 55.2 | <0.001* |
| | | Day 30 | 290.7 | 70.9 | * |
| | Hemoglobin (g/dl) | Day 7 | 15.3 | 2.4 | <0.001* |
| | Tremoglobin (g/ui) | Day 30 | 11.3 | 2.2 | * |
| (6) | Hematocrit (%) | Day 7 | 42.2 | 6.3 | <0.001* |
| <u> </u> | Tiematocrit (70) | Day 30 | 38.1 | 6.9 | * |
| | MCV (fl) | Day 7 | 97.3 | 8.2 | 0.002** |
| oq | We v (ii) | Day 30 | 90.3 | 8.5 | 0.002 |
| Placebo (n=100) | RDW (%) | Day 7 | 17.1 | 3.2 | 0.635 |
| | (/0) | Day 30 | 17.8 | 2.9 | |
| | Platelets (x1, 000/mm <sup>3</sup> ) | Day 7 | 178.3 | 100.3 | <0.001* |
| | Tatelets (XI, 000/IIIII) | Day 30 | 252.1 | 140.2 | * |
| | TLC $(x1, 000/mm^3)$ | Day 7 | 12.8 | 5.4 | <0.001* |
| | TLC (XI, UUU/IIIII ) | Day 30 | 17.4 | 8.1 | * |

Figure (10) Serum ferritin in lactoferrin group and placebo group

<sup>\*</sup> Statistically significant difference (p<0.05) \*\*Highly statistically significant difference (p<0.01).

Results



This figure shows that serum ferritin is significantly higher in lactoferrin group than the placebo group on day 30.

Figure (11) Hemoglobin level in both lactoferrin and placebo groups



This figure shows a serum hemoglobin is significantly higher in lactoferrin group than the placebo group on day 30.

Figure (12) Mean corpuscular volume value in both lactoferrin and placebo groups



MCV = Mean corpuscular volume

This figure shows a comparison of MCV level in both placebo and lactoferrin groups between day 7 and day 30. Being much higher in lactoferrin group than in placebo group on day 30.

Figure (13): Mean red cell distribution width (RDW) in both lactoferrin and placebo groups



This figure shows a comparison of RDW in both placebo and lactoferrin groups between day 7 and day 30. Being lower in lactoferrin group than in placebo group on day 30.

Figure (14): Mean hematocrit in both lactoferrin and placebo groups.



This figure shows a comparison of hematocrite level in both placebo and lactoferrin groups between day 7 and day 30. Being much higher in lactoferrin group than in placebo group on day 30.

Figure (15): Total leucocytic count (TLC) in both lactoferrin and placebo groups.



This figure shows a comparison of TLC in both placebo and lactoferrin groups between day 7 and day 30. Being lower in lactoferrin group than in placebo group on day 30.

Figure (16): Platelet count in both lactoferrin and placebo groups.



This figure shows a comparison of platelets in both placebo and lactoferrin groups between day 7 and day 30. No statistical difference was found between lactoferrin group and placebo group on day 7 and day 30.

Table(23): Weight gain in both study groups:

| Variable | Lactoferrin<br>(n=100) | Placebo<br>(n=100) | Test<br>value | P.<br>value |
|---|---|---|---|---|
| | Mean±SD | Mean±SD | | |
| Birth weight (kg) | 1.45±0.45 | 1.55±0.55 | 1.062 | 0.29 |
| Body weight on day 30 (kg) | 2.20±0.55 | 2.1±0.60 | 0.916 | 0.361 |
| Weight gain (kg) | 0.75±0.35 | 0.55±0.38 | 5.193 | 0.03* |

Independent samples T Test

This table shows that there was no significant statistical difference between birth weight and body weight on day 30.

Lactoferrin supplemented group showed significant statistical weight gain than placebo one.

<sup>\*</sup> Statistically significant difference (p<0.05)

<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

Figure(17): weight gain in both study groups.



This figure shows that the mean weight gain was higher in lactoferrin supplemented group than in placebo one.

Table (24): The need and frequency of blood transfusion.

| Variable | Lactoferrin (n=100) | Placebo<br>(n=100) | Test<br>value | P. value |
|---|---|---|---|---|
| | No.(%) | No.(%) | | |
| Need for blood transfusion | 0(0%) | 19(19%) | 18.84 | <0.001* |
| Frequency of blood transfusion | | | | |
| No blood transfusion | 100(100%) | 81(81%) | 18.54 | <0.001* |
| 1 transfusion | 0(0%) | 12(12%) | 10.72<br>7 | 0.001** |
| 2 transfusions | 0(0%) | 7(7%) | 5.329 | 0.021 |

Chi-square test

Highly statistically significant difference (p<0.01).

This table shows that there is no one in the lactoferrin group needed blood transfusion 0% while in placebo group 19 preterm (19%) needed blood transfusion with 7 preterm neonates (7) % for 2 transfusions.

<sup>\*</sup> Statistically significant difference (p<0.05

Figure (18): Need for blood transfusion in both study groups.



This figure shows the percentage of preterm neonates who needed blood transfusion in the 2 groups being nil in the lactoferrin supplemented group and 19 % in the placebo group.

Figure (19): Frequency of blood transfusion in both study groups.



This figure shows the percentage of frequency of blood transfusion in the 2 groups being nil in the lactoferrin supplemented group and 12 % and 7% in the placebo group needed once and twice blood transfusion respectively.

Table (25): Comparison between placebo and oral

| Radiology | | Placebo<br>group<br>(n=100) | | Lactoferrin<br>group<br>(n=100) | | Test<br>value | P.<br>value |
|---|---|---|---|---|---|---|---|
| | | No. | % | No. | % | | |
| Chast v. way | Free | 87 | 87.0 | 88 | 88.0 | 0.000 | 1.000 |
| Chest x ray | RDS | 13 | 13.0 | 12 | 12.0 | 0.000 | 1.000 |
| | Free | 27 | 27.0 | 22 | 22.0 | | |
| Abdominal x ray | NEC changes | 3 | 3.0 | 0 | 0.0 | 1.844 | 0.398 |
| | Not done | 70 | 70.0 | 78 | 78.0 | | |
| | Free | 22 | 22.0 | 0 | 0.0 | | |
| Pelviabdominal<br>Ultrasound | NEC changes | 3 | 3.0 | 0 | 0.0 | 1.844 | 0.398 |
| Omasound | Not done | 75 | 75.0 | 100 | 100.0 | | |

lactoferrin groups regarding chest x-ray , abdominal x ray and pelvi-abdominal Ultrasound.

Chi-square test

<sup>\*</sup> Statistically significant difference (p<0.05)

This table shows that there was non significant statistical difference between placebo and oral lactoferrin groups regarding chest x-ray , abdominal x ray and pelviabdominal ultrasound findings.

Figure (20): showing placebo and oral lactoferrin groups regarding chest X-ray, abdominal X-ray and pelvi-abdominal ultrasound.



<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

This figure show no stastical significant difference between placebo and oral lactoferrin supplemented group as regard chest X-ray, abdominal X-ray and pelviabdominal ultrasound.

Table (26): Comparison between placebo, and once daily lactoferrin supplemented groups as regard blood, CSF, stool, urine and fungal cultures.

| Cultures | | gr | cebo<br>oup<br>=100) | d:<br>gr | nce<br>ally<br>oup<br>=100) | Test<br>valu<br>e | P.<br>value |
|---|---|---|---|---|---|---|---|
| | | No<br>· | % | No<br>· | % | | |
| <b>Blood culture</b> | Positive cultures | 18 | 18.0 | 5 | 5.0 | 7.07 | 0.008* |
| | Negative | 82 | 82.0 | 95 | 95.0 | 4 | * |
| | Escherichia coli | 5 | 5.0 | 1 | 1.0 | 5.85 | 0.557 |
| | Staphylococcus aureus | 5 | 5.0 | 1 | 1.0 | 6 | |
| | Staphylococcus epidemidis | 3 | 3.0 | 1 | 1.0 | | |

| | Acinetobacter spp | 2 | 2.0 | 0 | 0.0 | | |
|---|---|---|---|---|---|---|---|
| | Klebseila | 1 | 1.0 | 1 | 1.0 | | |
| | Enterobacter cloacae | 1 | 1.0 | 0 | 0.0 | | |
| | Moraxella | 0 | 0.0 | 1 | 1.0 | | |
| | Pseudomonas | | | | | | |
| | aeruginosa | 1 | 1.0 | 0 | 0.0 | | |
| CSF culture | Negative or not done | 98 | 98.0 | 10<br>0 | 100 | 0.01 | 0.907 |
| | Escherichia coli | 2 | 2.0 | 0 | 0.0 | 4 | |
| G. L. | Negative or not done | 96 | 96.0 | 10<br>0 | 100 | 0.60 | |
| Stool culture | Escherichia coli | 3 | 3.0 | 0 | 0.0 | 8 | 0.748 |
| | Klebseila | 1 | 1.0 | 0 | 0.0 | | |
| Ilwino aultuma | Magativa or not dona | 10 | 100. | 10 | 100. | | |
| Urine culture | Negative or not done | 0 | 0 | 0 | 0 | 0.12 | 0.721 |
| Fungal blood | Nagativa or not dona | 10 | 100. | 10 | 100. | 8 | 0.721 |
| culture | Negative or not done | 0 | 0 | 0 | 0 | | |

Chi-square test

This table shows the positive and negative results of different cultures. Positive cultures are much lower of significant stastical value in the lactoferrin group than in the placebo one.

It shows that positive blood cultures affected by E.coli represent 27.7 % of the total positive blood cultures in the placebo group.

Staph.aureus shows 27.7 % positive in the total positive cultures in the placebo group.

E.coli and Staph.aureus represent the most common pathogens in the placebo group regarding positive blood cultures.

Table (27): Time needed to reach full feeding in days in placebo and oral lactoferrin supplemented groups.

| Data | Mean±SD | Placebo | Lactoferrin | Test value | P. value |
|------------|---------|-------------|-----------------|------------|----------|
| | | group n=100 | group n=100 | | |
| Time to | Mean±SD | 14.5±6.5 | 9.2±4. <b>0</b> | 6.867 | <0.001** |
| take full | | | | | |
| feeding in | | | | | |
| days | | | | | |

Independent samples T Testand Chi-square test,

<sup>\*</sup> Statistically significant difference (p<0.05)

<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

<sup>\*</sup> Statistically significant difference (p<0.05)

<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

This table shows that there is significant statistical value regarding time to reach full feeding in which that oral lacoferrin supplemented group has reached full feeding faster than placebo group.

Figure (21): Placebo and oral lactoferrin groups regarding time in days needed to reach full feeding.

Time to take full feeding in days



This figure shows the average time in days to reach full enteral feeding in both study groups. In the lacoferrin group the mean was  $9.2\pm4.0.SD$  days , while in the placebo group was  $14.5\pm6.5$  SD days.

## Table (28): Length of stay in the NICU in the two study groups.

| Variable | Lactoferrin<br>(n=100) | Placebo (n=100) | Test<br>value | P. value |
|---|---|---|---|---|
| | Mean±SD | Mean±SD | value | |
| Length of stay | 21.5±11.8 | 28.22±14.9 | 3.816 | <0.001* |

Test Independent samples T Test

Statistically significant difference (p<0.05) \*

The length of the hospital stay is much lower with significant value in the lactoferrin group than in the placebo one

<sup>.</sup>Highly statistically significant difference (p<0.01)\*\*

Figure (22):The length of the NICU stay in days in the two studied groups.



This figure shows that there is significant statistical value regarding the length of hospital stay in NICU which is much lower at the lactoferrin supplemented group than in the placebo one .

Table (29): Comparison between placebo group and once daily lactoferrin supplemented group as regards long term outcome:

| P. value | Test<br>value | Lacoferrin<br>group (n=100) | | Placebo group<br>(n=100) | | Long term output | | |
|---|---|---|---|---|---|---|---|---|
| value | value | % | .No | % | .No | | | |
| 1 000 | 0.0 | 0.0 | 0 | 1.0 | 1 | Positive | ROP | |
| 1.000 | 0.0 | 100.0 | 100 | 9.0 | 99 | Negative | KUI | |
| 1.000 | 0.0 | 2.0 | 2 | 1.0 | 1 | Positive | BPD | |
| 1.000 | 0.0 | 98.0 | 98 | 99.0 | 99 | Negative | DrD | |
| 0.082 1.354 | 0.0 | 0 | 3.0 | 3 | Positive | NEC | | |
| | 1.334 | 1.354 | 1.354 | 100 | 97.0 | 97 | Negative | NEC |

ROP= Retinopathy of prematurity ,BPD=

Bronchopulmonary dysplasia

NEC = necrotizing enterocolitis

Independent samples T Test and Chi-square test

\* Statistically significant difference (p<0.05)

This table shows that there was no significant statistical difference between placebo group and oral lactoferrin supplemented group as regard

retinopathy of prematurity , bronchopulmonary dysplasia and necrotizing enterocolitis.



<sup>\*\*</sup>Highly statistically significant difference (p<0.01).

### Figure(23): Long term outcome for placebo group .and oral lactoferrin group

Table (30) The number of preterm neonates which developed sepsis in both two studied groups.

| P. value | Once daily group (n=100) | | Placebo<br>(n=1 | | |
|---|---|---|---|---|---|
| | % | .No | % | .No | |
| **0.008 | 5.0 | 5 | 18.0 | 18 | Developed sepsis |

This table shows that there was 18 preterm neonates who developed sepsis in the placebo group in comparsion with 5 preterm neonates who developed sepsis in lactoferrin supplemented group .There is significant statistical value of development of sepsis being much lower in the lactoferrin supplemented group than the placebo one.

Table( 31): Fate after 1 month in the two study .groups

| P.<br>value | Placeb<br>o<br>(n=100 | Lactoferi<br>n (n=100) | | | |
|---|---|---|---|---|---|
| | 79 | 93 | No | Improved and discharged | |
| *0.009 | 79 | 93.0 | % | discharged | Fate after 1 |
| | 12 | 3 | No | Improved but still in | |
| | 12.0 | 3.0 | % | NICU | month |
| | 9 | 4 | No | | |
| | , | | | Died | |
| | 9.0 | 4.0 | % | | |

Chi-square test

Statistically significant difference (p<0.05) \*

This table shows the fate after one month in the 2 groups and it is significant for the lactoferrin group (P value = 0.009).

<sup>.</sup>Highly statistically significant difference (p<0.01)\*\*

Figure (24): Fate after one month in both studied groups.



This figure shows the fate in the 2 study groups after one month in the lactoferrin group 93 %of the preterm neonates were discharged in comparision with 79 % in the placebo group.3% of the lactoferrin group were improved but still in NICU in comparsion with 12% of the placebo group. While 4 % were died of the lactoferrin group and 9 % of the placebo one.

Table (32): Overall mortality in the study groups.

| | | | Lactoferin (n=100) | Placebo<br>(n=100) | P. value |
|---|---|---|---|---|---|
| Outcome | Compiesod | No. | 96 | 91 | 0.407 |
| | Survived | % | 96.0 | 91 | |
| | Died | No. | 4 | 9 | |
| | Died | % | 4.0 | 9.0 | |

Fisher exact test

This table shows the overall mortality of the 2 studied groups being non significant statistically.

<sup>\*</sup> Statistically significant difference (p<0.05) \*\*Highly statistically significant difference (p<0.01).